CLINICAL TRIAL: NCT07303426
Title: The Knowledge About the Underlying Cause of Hearing Loss in Children
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Anna Persson, PhD, Head of Development at the Hearing Habilitation Center for Children and Youth at Karolinska University Hospital, Karolinska Institutet
Other Study IDs: 2024-03470-01
Record Dates: First submitted 2025-12-05; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Hearing Loss
Keywords: childhood hearing loss; questionnaires; hearing loss aetiology
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Consists of children with bilateral sensorineural hearing loss and their care-givers
- Group B: Consists of both children and care-givers who answer forms anonymously.

SUMMARY:
This is a qualitative study to investigate children and their care-givers knowledge about the underlying aetiology of the childrens hearing loss. Both children and care-givers are given forms with questions about the type and level of hearing loss, if they know the cause and if it matters to them. This is to better understand the level of knowledge in both children and their care-givers about different causes of hearing loss. This will help to develop better clinical tools and routines of informing families about causal investigations in the future.

DETAILED DESCRIPTION:
The knowledge of the aetiology in children with sensorineural hearing loss - does it matter?

Introduction In Sweden, hearing screening of newborns, preschoolers and school children can detect hearing loss (HL) early in life. The prevalence of HL in high income countries is 1-2/1000 at birth, increases to 3-4/1000 in school children and around 5/1000 in children aged 15-18. In the Stockholm region, all children with HL in need of intervention are enrolled at the Hearing Habilitation for children and youth at Karolinska university hospital where they are followed up until they finish high school.

As finding out that your child has a hearing loss hearing loss can be quite difficult to understand and accept for parents, the timepoint of diagnosis is not always the most appropriate time to offer investigations of the cause of the hearing loss. However, there are no clinical guidelines as when to offer it. During the succeeding regular follow-up visits of children with HL at the Hearing habilitation it is a common clinical experience that few children know why they have a HL and how it may change over their life course, and when they ask their parents, they do not know either. A reason for this may be that some parents were informed when their child was diagnosed years ago and chose not to investigate the cause. Another comment from parents, in cases where many years have passed since the diagnosis, is that some parents do not remember if they received a question about investigating the cause or not. This give rise to an ethical question from the child´s point of view; should the audiology doctor ask the parents if they want to investigate the cause of the HL again, or should they ask the child themselves? With age, children themselves may wonder: what is the cause of my HL and how will that affect my future? The knowledge and interest around the cause of the hearing loss is something that has not been investigated in a systematic manner before, but is important to provide the child with HL and their parents with the right support in the right time. As some etiologies affect other areas of development, knowing about the etiology of the hearing loss also gives professionals cues to provide the most optimal intervention. In this study, we want to examine what the caregivers of children as well as the children themselves know and how important they think it is to know about the cause of HL. Another motivation to pursue this study is that we do not know how many children in the intended target group who have investigated the etiology.

Scientific questions:

1. Do caregivers and children with HL know the cause of the child's HL?
2. What difference does knowing/not knowing about the cause of HL make for the children themselves and their parents?
3. Do caregivers and children have different opinions about the importance of investigating the cause of HL?

Study design To collect data we will use a patient-related outcome measure (PROM) with questions specifically made for this study together with information around background variables. Information about the study and consent form will be mailed out to all children/youth enrolled at the Hearing Habilitation for Children and Youth born between 2010-2015 with diagnosis code H90.3 (bilateral sensorineural hearing loss) (n=327) and their guardians.

Procedures and materials

1. Children with different types and degrees of HL born 2010-2015 and their parents enrolled at the Hearing Habilitation. Recruitment via letter home with information about the study, consent form and prepaid return envelope followed by a letter with a QR code/paper version.
2. Children/families will be invited to complete a questionnaire (digital or/paper version) separately (questions about their knowledge about the cause of hearing loss) and a background form filled in by the child's parents (age, sex, type and degree of HL).

Clinical implications This project is one of the first to investigate this important, yet, challenging part of the intervention in children. In the Swedish healthcare system, children are supposed to seek help themselves from 13 years of age. As there is no systematically collected information on group level around the knowledge of the cause of hearing loss in this target group, the results from this study may contribute to a better understanding as to the importance of etiological diagnosis and surveillance of each child with HL. It will also act as a guidance to medical professionals and families to better understand the cause of HL and expectations of the child's hearing, speech and language development.

ELIGIBILITY:
Inclusion Criteria:

* Children with Hearing loss and their care-givers

Exclusion Criteria:

* Children with no hearing loss or care-givers to children with no hearing loss.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with hearing loss and their care-givers
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2024-09-09 (Actual); Primary Completion 2025-05-22 (Actual); Study Completion 2025-05-22 (Actual)

PRIMARY OUTCOMES:
Do caregivers and children with HL know the cause of the child's HL | from sept 2024 to may 2025
  To study weather children and care-givers know the cause of the childs HL if available.
To investigate children´s and caregivers perspectives on the importance of knowing the cause of the child´s hearing loss through questionnaires. | Group A: Sept 2024 to Nov 2024, Group B: Jan 2025 to May 2025
  Questionnaires were distrubuted wither through mail or QR code for the parents and children to respond.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Universitetssjukhuset, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No
IPD is only for this study